CLINICAL TRIAL: NCT04400903
Title: A Prospective, Multi-Center Investigational Study of Heart Rate Variability Monitoring for the Early Detection of Pancreatic Cancer
Brief Title: Monitoring Heart Rate Variability for the Early Detection of Pancreatic Cancer
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); American Association for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aaron Grossberg, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00021185; NCI-2020-03178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021185 (Other: OHSU Knight Cancer Institute); R01CA264133 (NIH)
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Stage I Pancreatic Cancer AJCC v8; Stage IA Pancreatic Cancer AJCC v8; Stage IB Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (HRV monitoring, questionnaire): Participants undergo HRV monitoring using an activity monitor (WHOOP) for a minimum of 5 days weekly for up to 1 year in patients with newly-diagnosed PDAC and up to 5 years for patients in high risk group.
  Interventions: Device: Activity Monitor; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Device: Activity Monitor — Undergo HRV monitoring via WHOOP device
  Other Names: Activity Tracker; Activity Tracker Device; Physical Activity Measuring Device
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines heart rate monitoring variability for the early detection of pancreatic cancer. Pancreatic cancer is a very difficult disease to detect early. This study is being done to observe the heart rate variability in patients with pancreatic cancer compared to undiagnosed individuals with increased risk of developing pancreatic cancer. This may help researchers determine if pancreatic occurrences/recurrences (chance of coming back) can be detected sooner through monitoring heart rate and activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether heart rate variability (HRV) is reduced in patients with pancreatic ductal adenocarcinoma (PDAC) compared with individuals at increased risk of developing PDAC. (Stage I) II. To assess the feasibility of long-term compliance using a wearable device. (Stage II)

SECONDARY OBJECTIVES:

I. To assess compliance with using a wearable device. (Stage I and II) II. To validate effectiveness of virtual device training. (Stage I and II) III. To determine whether HRV is reduced in participants at high-risk of developing PDAC. (Stage II) IV. To characterize timing and occurrence of PDAC among high-risk without disease. (Stage II) V. To characterize timing and occurrence of PDAC among participants at high-risk of developing PDAC. (Stage II)

EXPLORATORY OBJECTIVES:

I. To investigate the relationship between changes in HRV relative to sarcopenia-related body composition characteristics in PDAC patients. (Stage I) II. To investigate the relationship between the pNN50 HRV measure and PDAC diagnosis. (Stage I and II) III. To compare changes in sleep biometrics among all participants. (Stage I and II) IV. To evaluate changes in health-related quality of life assessments among all participants. (Stage I and II) V. To evaluate participant satisfaction with virtual device instruction.

OUTLINE:

Participants undergo HRV monitoring using an activity monitor (WHOOP) for a minimum of 5 days weekly for up to 1 year in patients with newly-diagnosed PDAC and up to 5 years for patients in high risk group.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign an informed consent document
* Own a smartphone that uses Android or Apple iOS operating systems
* Participant must have one of the following:

  * Individuals with newly-diagnosed, treatment naive PDAC - all stages (applicable to Stage 1 only), or
  * Individuals with at least one of the following family phenotype and age will be included:

    * Two or more relatives with PDAC on the same side of the family, where 2 PDAC affected individuals are first-degree related (FDR) AND at least one PDAC-affected individual is an FDR of the subject; Age >= 50 years OR 10 years before onset in family
    * Two affected FDR with PDAC; Age >= 50 years OR 10 years before onset of an FDR
    * Any of BRCA1, BRCA2, PALB2, ATM mutations confirmed pathogenic or likely pathogenic; Age >= 50 years OR 10 years before onset of an FDR or second-degree relative (SDR)
    * Familial atypical multiple mole-melanoma (FAMMM) with confirmed pathogenic or likely pathogenic mutation variants in: p16, CDKN2A; Age >= 50 years
    * Known mutation carrier for STK11 (Peutz-Jeghers syndrome); Age >= 50 years
    * Lynch syndrome (hereditary nonpolyposis colorectal cancer [HNPCC]) with confirmed pathogenic or likely pathogenic variants in: MLH1, MSH2, MSH6, PMS2, or EPCAM; Age >= 50 years OR 10 years before onset of an FDR or SDR
    * Hereditary pancreatitis with confirmed PRSS1 pathogenic or likely pathogenic history of pancreatitis; Age >= 50 years

Exclusion Criteria:

* Any medical conditions that in the opinion of the investigators would compromise participant safety and/or the integrity of the data

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PDAC and participants at high risk for PDAC at Oregon Health and Science University, New York University and University of Nebraska Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Magnitude of heart rate variability (HRV) decline (Stage I) | Up to 1 year after enrollment
  As measured by root mean square of the successive differences (RMSSD) in pancreatic ductal adenocarcinoma (PDAC) patients and in high-risk participants.
Compliance statistics for wristband use (Stage II) | Until onset of PDAC, study withdrawal, or death, whichever occurs first, assessed up to 5 years after enrollment
  Defined as the percentage of days during which data were collected during at least 70% of the hours.

SECONDARY OUTCOMES:
Compliance statistics for wristband use for all participants (Stage I, II) | Up to 6 weeks and 6 months after enrollment and device activation
  Defined as the percentage of days during which data were collected for at least 70% of the hours.
Effectiveness of virtual training (Stage I, II) | Up to 1 week after enrollment and device activation
  Defined as the percentage of participants for whom high quality data are available within 3 days of set up. The pattern of missing data, and the percentage of participants able to collect data will be presented graphically. Will also associate the compliance with patient characteristics, regions and seasons to understand what may impact the compliance rate.
Magnitude of HRV change (Stage II) | Up to 5 years post enrollment
  As measured by RMSSD, in participants at high-risk of developing PDAC.
Incidence of PDAC among high-risk participants (Stage II) | Up to 5 years post enrollment
Time of PDAC diagnosis among high-risk participants who developed PDAC (Stage II) | Up to 5 years post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Grossberg, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - OHSU Knight Cancer Institute, Portland, Oregon